CLINICAL TRIAL: NCT03201237
Title: Main Researcher for Action Observation Training (AOT)
Brief Title: Comparison of Short- and Long-time Action Observation Training on Upper Limb Function in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Do hyun Kim, Principal Investigator for AOT, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InjeU3
Record Dates: First submitted 2017-06-20; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 min AOT (Experimental)
  Interventions: Other: Action observation training
- 60 min AOT (Placebo Comparator)
  Interventions: Other: Action observation training

INTERVENTIONS:
Other: Action observation training — Each child observed a task video and then performed a task

SUMMARY:
To compared short- and long-time action observation training (AOT) in terms of grip strength, the Jebsen Taylor Hand Function Test (JTHF), the Quality of Upper Extremities Skills Test (QUEST), and the ABILHAND-Kids test.

ELIGIBILITY:
Inclusion Criteria:

* ages between 6 and 15 years
* confirmed diagnosis of spastic CP
* below grade 2 on the modified Ashworth scale
* between grade 4 and 8 on the house functional classification system
* ability to understand the assessor's instructions.

Exclusion Criteria:

* severe spasticity in UL (MAS>2)
* orthopedic surgery in the UL within 6 months
* absence of sensory

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change of grip strength | 6 months
  Power of hand grip

CONTACTS AND LOCATIONS:
Overall Officials: Do H Kim, MS, Principal Investigator — Inje University
Locations (1):
- Inje University, Gimhae, Gyeongsangnam-do, South Korea